CLINICAL TRIAL: NCT05300191
Title: In Vitro Analysis of Effluent Dialysate Solution From Patients on Peritoneal Dialysis, With the CloudCath Device
Status: Suspended | Type: Observational
Why Stopped: temporary pause due to business priorities
Sponsor: CloudCath (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-L-003
Record Dates: First submitted 2022-03-09; First posted 2022-03-29 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Peritoneal Dialysis-associated Peritonitis; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Peritoneal dialysis patients: Patients undergoing peritoneal dialysis. Patients may be using either Continuous Ambulatory Peritoneal Dialysis (CAPD), Continuous Cycling Peritoneal Dialysis (CCPD) or Intermittent Peritoneal Dialysis (IPD).
  Interventions: Diagnostic Test: Effluent dialysate

INTERVENTIONS:
Diagnostic Test: Effluent dialysate — Effluent dialysate samples evaluated for evidence of peritonitis

SUMMARY:
A proof-of-concept study of a prototype CloudCath device designed to detect peritonitis using the effluent dialysate from patients undergoing peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females with end-stage renal disease on peritoneal dialysis for a minimum of 10 days prior to obtaining the specimen.
* Specimens shall be leftover (or remnant) from a specimen that has been drained as part of the routine care for the patient.
* Specimens shall not contain any individually identifiable information from the patient it was obtained from.

Exclusion Criteria:

* Patients providing specimens should not be under the administration of any antibiotics other than those utilized for the treatment of peritonitis.
* Patients providing specimens should not suffer from a known liver disease or from ovarian or liver cancer.
* Patients providing specimens should not be under the administration of calcium channel blockers or amlodipine for less than 30 days prior to providing a specimen.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients currently using peritoneal dialysis and at elevated risk for developing peritonitis.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Spectral measurements of effluent dialysate solutions | immediately post dialysis
  a quantitative analysis of the spectral characteristics of the effluent dialysate solution using a proprietary algorithm and sensing equipment that results in a quantitative CloudCath Score.
Conductivity measurements of effluent dialysate solutions. | immediately post dialysis
  a quantitative assessment of conductivity of the effluent dialysate solution using a proprietary algorithm and sensing equipment that results in a quantitative CloudCath Score.

CONTACTS AND LOCATIONS:
Overall Officials: Ben Briggs, MD, PhD, Study Director — University of California, San Francisco
Locations (1):
- CloudCath Investigational Site, Guadalajara, Jalisco, Mexico